CLINICAL TRIAL: NCT05443724
Title: A 52-week, Phase 2, Open-label Trial to Evaluate the Long-term Safety and Tolerability of CVL-231 (Emraclidine) in Adult Participants With Schizophrenia
Brief Title: A Study to Evaluate Safety and Tolerability of CVL-231 (Emraclidine) in Adult Participants With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVL-231-2003; 2022-001151-16 (EudraCT Number)
Record Dates: First submitted 2022-06-29; First posted 2022-07-05 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Schizophrenia
Keywords: Schizophrenia Spectrum and Other Psychotic Disorders; Mental Disorders
MeSH Terms: conditions — Schizophrenia; Schizophrenia Spectrum and Other Psychotic Disorders; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CVL-231 30 mg (Experimental): Participants will receive CVL-231 30 milligrams (mg) tablet, once daily for 52 weeks.
  Interventions: Drug: CVL-231 30 mg

INTERVENTIONS:
Drug: CVL-231 30 mg — Oral tablets
  Other Names: Emraclidine

SUMMARY:
The primary purpose of this study is to assess the long-term safety and tolerability of oral emraclidine in adult participants with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

1. Completed 6 weeks of post-randomization treatment in Trial CVL-231-2001 (NCT05227690) or CVL-231-2002 (NCT05227703) and who, in the opinion of the investigator, could potentially benefit from treatment with emraclidine for schizophrenia.
2. Primary diagnosis of schizophrenia per Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5), as confirmed by the Mini International Neuropsychiatric Interview (MINI) for Psychotic Disorders.
3. Participants who have been stable on antipsychotic medication for at least one 3-month in the year prior to screening.
4. Outpatient status at the time of signing the informed consent form informed consent form (ICF).
5. Willing to discontinue all prohibited medications to meet protocol-required washouts prior to and during the trial period.
6. Ability, in the investigator's opinion, to understand the nature of the trial, participate in trial visits, and comply with protocol requirements.

Exclusion Criteria:

1. Current DSM-5 diagnosis other than schizophrenia (note: anxiety symptoms secondary to schizophrenia are allowed.

   * Acute depressive symptoms within 30 days prior to signing the ICF that require treatment with an antidepressant are exclusory.
   * Acute manic symptoms within 30 days prior to signing the ICF that require treatment with a mood stabilizer are exclusory.
2. Any of the following:

   * Schizophrenia is considered resistant/refractory to antipsychotic treatment by history (failure to respond to 2 or more courses of adequate pharmacological treatment defined as an adequate dose per label and a treatment duration of at least 4 weeks).
   * History of response to clozapine treatment only or failure to respond to clozapine treatment.
3. Current or past history of significant cardiovascular, pulmonary, gastrointestinal, renal, hepatic, metabolic, genitourinary, endocrine (including diabetes mellitus), malignancy (except for basal cell carcinoma of the skin and cervical carcinoma in situ, at the discretion of the investigator), hematological, immunological, neurological, or psychiatric disease that, in the opinion of the investigator or medical monitor, could compromise either participant safety or the results of the trial.
4. Active central nervous system infection, demyelinating disease, degenerative neurological disease, brain tumor, prior hospitalization for severe head trauma, seizures (excluding febrile seizures in childhood), or any central nervous system disease deemed to be progressive during the trial that may confound the interpretation of the trial results
5. Diagnosis of moderate to severe substance or alcohol use disorder (excluding nicotine or caffeine) as per DSM-5 criteria within 12 months prior to signing the ICF.
6. Risk for suicidal behavior as assessed by the C-SSRS and investigator's clinical assessment.
7. Any condition that could possibly affect drug absorption, including, but not limited to bowel resections, bariatric weight loss surgery, gastric banding, and gastrectomy
8. Use of prohibited medications prior to randomization within the required wash-out period or likely to require prohibited concomitant therapy during the trial.
9. Clinically significant abnormal findings on the physical examination, medical history review, ECG, or clinical laboratory results at screening.
10. Positive pregnancy test result prior to receiving investigational medicinal product (IMP).

Note: female participants who are pregnant, breastfeeding, or planning to become pregnant during IMP treatment or within 7 days after the last dose of the IMP are also excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2022-09-02 (Actual); Primary Completion 2025-06-25 (Actual); Study Completion 2025-06-25 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment Emergent Adverse Events (TEAEs) | Up to Week 56
Number of Participants With Clinically Significant Changes in Vital Sign Values | Up to Week 52
Number of Participants With Clinically Significant Changes in Body Weight | Up to Week 52
Number of Participants With Clinically Significant Changes in Physical and Neurological Examination Results | Up to Week 52
Number of Participants With Clinically Significant Changes in Electrocardiogram (ECG) Values | Up to Week 52
Number of Participants With Clinically Significant Changes in Clinical Laboratory Values | Up to Week 52
Number of Participants With Clinically Significant Changes in Metabolic Parameter Values | Up to Week 52
Number of Participants With Clinically Significant Change in Columbia Suicide Severity Rating Scale (C-SSRS) Score | Up to Week 52
Number of Participants With Change from Baseline in Extrapyramidal Symptoms Measured by the Simpson Angus Scale (SAS) Score | Baseline up to Week 52
Number of Participants With Change from Baseline in Extrapyramidal Symptoms Measured by the Abnormal Involuntary Movement Scale (AIMS) Score | Baseline up to Week 52
Number of Participants With Change from Baseline in Extrapyramidal Symptoms Measured by the Barnes Akathisia Rating Scale (BARS) Score | Baseline up to Week 52

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (66):
- United States (49):
  - Phoenix, Arizona, Phoenix, Arizona
  - Bryant, Arkansas, Bryant, Arkansas
  - Little Rock, Arkansas, Little Rock, Arkansas
  - Anaheim, California, Anaheim, California
  - Bellflower, California, Bellflower, California
  - Culver City, California, Culver City, California
  - Garden Grove, California, Garden Grove, California
  - La Habra, California, La Habra, California
  - Lemon Grove, California, Lemon Grove, California
  - Montclair, California, Montclair, California
  - Orange,California, Orange, California
  - Pico Rivera, California, Pico Rivera, California
  - Riverside, California, Riverside, California
  - San Diego, California, San Diego, California
  - Sherman Oaks, California, Sherman Oaks, California
  - Torrance, California, Torrance, California
  - Walnut Creek, California, Walnut Creek, California
  - New Haven, Connecticut, New Haven, Connecticut
  - Bonita Springs,Florida, Bonita Springs, Florida
  - Fort Myers, Florida, Fort Myers, Florida
  - Hialeah, Florida, Hialeah, Florida
  - Miami, Florida, Miami, Florida
  - Miami Lakes, Florida, Miami Lakes, Florida
  - Miami Springs, Florida, Miami Springs, Florida
  - Oakland Park, Florida, Oakland Park, Florida
  - West Palm Beach, Florida, West Palm Beach, Florida
  - Atlanta, Georgia, Atlanta, Georgia
  - Decatur, Georgia, Decatur, Georgia
  - Savannah,Georgia, Savannah, Georgia
  - Berwyn, Illinois, Berwyn, Illinois
  - Chicago, Illinois, Chicago, Illinois
  - Marrero, Louisiana, Marrero, Louisiana
  - Shreveport, Louisiana, Shreveport, Louisiana
  - Gaithersburg, Maryland, Gaithersburg, Maryland
  - Flowood, Mississippi, Flowood, Mississippi
  - Las Vegas, Nevada, Las Vegas, Nevada
  - Berlin, New Jersey, Berlin, New Jersey
  - Cedarhurst, New York, Cedarhurst, New York
  - New York, New York, New York, New York
  - Staten Island, New York, Staten Island, New York
  - Charlotte, North Carolina, Charlotte, North Carolina
  - North Canton, Ohio, North Canton, Ohio
  - Oklahoma City, Oklahoma, Oklahoma City, Oklahoma
  - Franklin,Tennessee, Franklin, Tennessee
  - Austin, Texas, Austin, Texas
  - DeSoto, Texas, DeSoto, Texas
  - Houston, Texas, Houston, Texas
  - Plano, Texas, Plano, Texas
  - Richardson, Texas, Richardson, Texas
- Bulgaria (8):
  - Sofia, Sofia-Grad, Sofia, Sofia-Grad
  - Pazardzhik, Pazardzhik, Pazardzhik
  - Pleven, Pleven, Pleven
  - Sliven, Sliven, Sliven
  - Stara Zagora, Stara Zagora, Stara Zagora
  - Varna, Varna, Varna
  - Veliko Tarnovo, Veliko Tarnovo, Veliko Tarnovo
  - Vratsa, Vratsa, Vratsa
- Hungary (2):
  - Kalocsa, Bács-Kiskun, Kalocsa, Bács-Kiskun county
  - Gyor, Gyor-Moson-Sopron, Győr, Győr-Moson-Sopron
- San Juan, Puerto Rico, San Juan, Puerto Rico
- Ukraine (6):
  - Ivano Frankivsk, Ivano Frankivsk, Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Lviv, L'vivs'ka Oblast, Lviv, Lviv Oblast
  - Kropyvnytskyi, Kropyvnytskyi, Kropyvnytskyi
  - Kyiv, Kyïv, Kyiv
  - Smila, Smila, Smila
  - Vinnytsia, Vinnytsia, Vinnytsia

IPD SHARING:
Plan to Share IPD: No